CLINICAL TRIAL: NCT06442215
Title: Selection of Surgical Technique in Rectal Cancer Through the Development of a Predictive Model for Optimal Oncological Outcomes
Brief Title: Selection of Surgical Technique in Rectal Cancer
Acronym: TECARE
Status: Recruiting | Type: Observational
Sponsor: Institut d'Investigació Biomèdica de Girona Dr. Josep Trueta (Other)
Responsible Party: Sponsor
Other Study IDs: 2024.017
Record Dates: First submitted 2024-05-29; First posted 2024-06-04 (Actual); Last update posted 2024-06-05 (Actual); Status verified 2024-06

CONDITIONS: Rectal Neoplasms
Keywords: Rectal cancer; Surgery; Minimal invasive surgery; Oncological outcomes
MeSH Terms: conditions — Rectal Neoplasms | interventions — Data Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients undergoing elective surgery for rectal neoplasm: Patients diagnosed with rectal neoplasia undergoing elective surgery between 2017 and 2021 at medical centers within the national territory.
  Interventions: Other: Data collection

INTERVENTIONS:
Other: Data collection — Collection of preoperative demographic, clinical, and radiological variables from patients who meet the inclusion criteria in order to identify possible risk factors for suboptimal surgical treatment

SUMMARY:
Currently, there is no prediction scale available to identify patients with rectal neoplasms as technically complex in the middle and lower thirds; that is, those who are at high risk of affected circumferential margins and low quality of the mesorectum. The application of a predictive model that allows preoperative identification of the group of patients in whom optimal results in mesorectal quality and circumferential margin are less likely to be obtained through laparoscopic or minimally invasive surgery would enable the selection of patients who will require and justify all efforts and healthcare resources to improve surgical outcomes.

Therefore, the investigators aim to create a predictive model to identify these patients, allowing the discrimination of which patients will benefit from different techniques, or even which ones would be opportune to initially consider an open approach.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled surgery for anterior resection of the rectum meeting oncological criteria with mesorectal excision.
* Age ≥ 18 years.
* Histology of adenocarcinoma with or without neoadjuvant chemotherapy or chemoradiotherapy.
* Initial stage T1-T4a. Any N. Any M.
* Intention for R0 resection.

Exclusion Criteria:

* Colorectal tumor with histology different from adenocarcinoma.
* Synchronous colon tumor.
* Benign pathology or adenoma.
* Tis.
* T4b or oncological multivisceral resections.
* History of neoplastic colorectal surgery or local excision or TAMIS.
* Perforated or obstructive rectal neoplasm.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with rectal neoplasia undergoing elective surgery during a period of time from 2017 to 2021
Sampling Method: Non-Probability Sample
Enrollment: 333 (Estimated)
Dates: Start 2024-04-03 (Actual); Primary Completion 2025-04-03 (Estimated); Study Completion 2026-04-03 (Estimated)

PRIMARY OUTCOMES:
Suboptimal oncological outcomes | 15 postoperative days
  Surgical resection with affected margins (proximal-distal and/or circumferential < 1mm) and/or incomplete or nearly complete mesorectal resection

SECONDARY OUTCOMES:
Surgical and Postoperative complications | 30 postoperative days
  Conversion to open surgery and anastomotic dehiscence rates
Overall and disease free survival | 3-years surgery
  Recurrence of the tumoral disease at the pelvic level and distant recurrence is defined as s the recurrence of the disease in other distant organs.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitari Dr. Josep Trueta de Girona, Girona, Spain

IPD SHARING:
Plan to Share IPD: No